CLINICAL TRIAL: NCT03720132
Title: Optimization of Therapeutic Drug Monitoring of Vancomycin in Pediatric Patients With an Implanted Port Catheter
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Emerging evidence made the trial unnecessary.
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Isabelle Spriet, PharmD, PhD, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S20140519
Record Dates: First submitted 2016-11-29; First posted 2018-10-25 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Catheter Related Blood Stream Infections
Keywords: Vancomycin; Therapeutic drug monitoring; Catheter related blood stream infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with port catheter: flushing (Experimental): In patients with a catheter-related blood stream infection (CRBSI) and a port catheter, being treated with vancomycin intravenously, we will flush the catheter with 30 ml of sodium chloride 0.9 % prior to blood sampling to determine vancomycin concentrations, in order to decrease residuel vancomycin in the port.
  Interventions: Procedure: Extensive flushing of the port catheter

INTERVENTIONS:
Procedure: Extensive flushing of the port catheter — The port catheter will be flushed extensively with sodium chloride 0.9% before blood sampling. Blood sampling will occur through the central catheter and peripherally simultaneously.

SUMMARY:
The goal of this study is to verify whether extensive flushing of the port catheter in patients with catheter related blood stream infection will lead to correct vancomycin trough levels, taken via the port catheter and compared with simultaneously taken peripheral samples.

DETAILED DESCRIPTION:
In this study, extensive flushing of the port catheter prior to blood sampling to determine vancomycin trough levels, will be compared with normal flushing. To ascertain correctness of the trough levels taken via the central catheter, sampling will occur through a peripheral catheter simultaneously.

Flushing will be done with sodium chloride 0.9 % solution.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with a port catheter
* Treated with systemic vancomycin and/or vancomycin "lock"

Exclusion Criteria:

* Age > 18 years
* Active downgrading of care

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Vancomycin trough levels via port catheter and peripheral vein | At steady state i.e. approximately 36 hours after initation of the treatment or a change in dose
  Vancomycin trough levels will be determined, both on peripheral blood and blood taken via the port catheter and will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PharmD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

REFERENCES:
- [Background] Rybak MJ, Lomaestro BM, Rotschafer JC, Moellering RC, Craig WA, Billeter M, Dalovisio JR, Levine DP. Vancomycin therapeutic guidelines: a summary of consensus recommendations from the infectious diseases Society of America, the American Society of Health-System Pharmacists, and the Society of Infectious Diseases Pharmacists. Clin Infect Dis. 2009 Aug 1;49(3):325-7. doi: 10.1086/600877. PMID 19569969
- [Background] Wright DF, Al-Sallami HS, Jackson PM, Reith DM. Falsely elevated vancomycin plasma concentrations sampled from central venous implantable catheters (portacaths). Br J Clin Pharmacol. 2010 Nov;70(5):769-72. doi: 10.1111/j.1365-2125.2010.03749.x. No abstract available. PMID 21039771
- [Background] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710